CLINICAL TRIAL: NCT01653795
Title: A Randomized Trial Comparing the Laryngeal Mask Airway-Unique and Laryngeal Mask Airway-Supreme in Children
Brief Title: A Comparison of the Laryngeal Mask Airway (LMA) - Unique and LMA-Supreme in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Narasimhan Jagannathan, Principal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: LMA-U vs SLMA (multiple sizes)
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Laryngeal Mask Airway in Children
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LMA Unique (Active Comparator)
  Interventions: Device: LMA Unique: control device
- LMA Supreme (Active Comparator)
  Interventions: Device: LMA Supreme: comparison device

INTERVENTIONS:
Device: LMA Unique: control device — LMA Unique will be placed in children based on a computer generated randomization. One of four different sizes of airways will be used: 1.5, 2.0, or 2.5. The size of the airway device will be determined according to the manufacturer's guidelines that are standardized by the patient's weight in kilograms.
  Other Names: Laryngeal Mask Airway
  Arms: LMA Unique
Device: LMA Supreme: comparison device — LMA Supreme will be placed in children based on a computer generated randomization. One of four different sizes of airways will be used: 1.5, 2.0, or 2.5, The size of the airway device will be determined according to the manufacturer's guidelines that are standardized by the patient's weight in kilograms.
  Other Names: Laryngeal Mask Airway
  Arms: LMA Supreme

SUMMARY:
The aim of this randomized prospective study is to compare two single-use laryngeal mask airways the LMA Unique and the LMA Supreme, in pediatric patients. The investigators hypothesize that airway leak pressures with the LMA Supreme will be superior to the LMA Unique.

DETAILED DESCRIPTION:
The goal of this study is to compare the LMA Unique and LMA-Supreme in children undergoing anesthesia. The investigators hypothesize that airway leak pressures with the LMA Supreme will be superior when compared with the LMA Unique at two different standardized intracuff pressures (40 and 60 cm H20). Airway leak pressures will be measured by recording the circuit pressure at which equilibrium is reached. The ease of placement, fiberoptic grade of laryngeal view, feasibility of use, and complications will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing general anesthesia using a supraglottic airway device

Exclusion Criteria:

* ASA class IV, V, Emergency procedures
* active respiratory infection
* known history of difficult mask ventilation
* a diagnosis of a congenital syndrome associated with difficult airway management
* airway abnormalities (e.g., laryngomalacia, subglottic stenosis)
* active gastrointestinal reflux
* coagulopathy
* clinically significant pulmonary disease(s)

Ages: 3 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Airway Leak Pressure | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Airway leak pressures will be measured by recording the circuit pressure at which equilibrium is reached when fresh gas flow is delivered at 3L/min when the pressure limiting valve is closed.

SECONDARY OUTCOMES:
Time to secure the airway | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  From picking up the airway device to bilateral chest expansion and presence of ETCO2
Number of attempts to place the device | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Number of attempts needed for successful placement will be recorded (maximum of 3 attempts will be considered as a failure)
Fiberoptic grade of laryngeal view | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The laryngeal alignment through the devices will be graded using an established scoring system
Gastric insufflation | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The presence of gastric insufflations will be assessed during leak pressure testing by using epigastric auscultation
Ease of gastric tube placement (only in patients who receive LMA Supreme) | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The ease of gastric placement will be timed and assessed using a subjective scale. The LMA Unique does not contain a gastric port so this outcome will only be assessed in patients who received the LMA Supreme device.
Quality of the airway | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The quality of hands free anesthesia will be assessed during maintenance of anesthesia using a previously described scale
Incidence of device repositioning and/or replacement | Participants will be followed for the duration of anesthesia and after surgery, an average of 24 hours
  Intra-operative device repositioning or replacement of the device due to excessive air leak or airway obstruction, as evidenced by an obstructive pattern on the continuous end-tidal carbon dioxide monitor that leads to a decrease in oxygen saturation by pulse oximetry to less than 90%.
Oropharyngolaryngeal morbidity at discharge | Participants will be followed for the duration of anesthesia and after surgery, an average of 24 hours
  Assessed by the subject's response or parents subjective assessment to standardized questions regarding oropharyngeal complaints such as sore throat, jaw pain, neck discomfort.
Oropharyngolaryngeal morbidity at 24 hours post-operatively | Measured at 24 hours after device placement/study initiation
  Assessed by the subject's response or parents subjective assessment to standardized questions regarding oropharyngeal complaints such as sore throat, jaw pain, neck discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Narasimhan Jagannathan, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Jagannathan N, Sohn LE, Sawardekar A, Gordon J, Langen KE, Anderson K. A randomised comparison of the LMA SupremeTM and LMAProSealTM in children. Anaesthesia. 2012 Jun;67(6):632-9. doi: 10.1111/j.1365-2044.2012.07088.x. Epub 2012 Mar 15. PMID 22420717
- [Background] Jagannathan N, Sohn LE, Chang E, Sawardekar A. A cohort evaluation of the laryngeal mask airway-Supreme in children. Paediatr Anaesth. 2012 Aug;22(8):759-64. doi: 10.1111/j.1460-9592.2012.03832.x. Epub 2012 Mar 15. PMID 22416790
- [Background] Jagannathan N, Sohn LE, Sawardekar A, Chang E, Langen KE, Anderson K. A randomised trial comparing the laryngeal mask airway Supreme with the laryngeal mask airway Unique in children. Anaesthesia. 2012 Feb;67(2):139-44. doi: 10.1111/j.1365-2044.2011.06960.x. Epub 2011 Nov 9. PMID 22070630
- [Background] Lee JR, Kim MS, Kim JT, Byon HJ, Park YH, Kim HS, Kim CS. A randomised trial comparing the i-gel (TM) with the LMA Classic (TM) in children. Anaesthesia. 2012 Jun;67(6):606-11. doi: 10.1111/j.1365-2044.2012.07072.x. Epub 2012 Feb 21. PMID 22352745
- [Background] Goyal R, Shukla RN, Kumar G. Comparison of size 2 i-gel supraglottic airway with LMA-ProSeal and LMA-Classic in spontaneously breathing children undergoing elective surgery. Paediatr Anaesth. 2012 Apr;22(4):355-9. doi: 10.1111/j.1460-9592.2011.03757.x. Epub 2011 Dec 8. PMID 22151106
- [Background] Beringer RM, Kelly F, Cook TM, Nolan J, Hardy R, Simpson T, White MC. A cohort evaluation of the paediatric i-gel() airway during anaesthesia in 120 children. Anaesthesia. 2011 Dec;66(12):1121-6. doi: 10.1111/j.1365-2044.2011.06884.x. Epub 2011 Sep 1. PMID 21883132